CLINICAL TRIAL: NCT04550520
Title: Copeptin After a Subcutaneous Stimulation With Glucagon in Adults (Healthy Volunteers and Patients With Diabetes Insipidus or Primary Polydipsia) - The Glucacop-Study
Brief Title: Copeptin After a Subcutaneous Stimulation With Glucagon in Adults
Acronym: Glucacop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2020-02038; me20ChristCrain
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Insipidus
Keywords: Copeptin; Glucagon; central diabetes insipidus; primary polydipsia; hypothalamo-pituitary-adrenal axis; posterior pituitary gland; polyuria-polydipsia syndrome
MeSH Terms: conditions — Diabetes Insipidus; Diabetes Insipidus, Neurogenic; Polydipsia, Psychogenic

STUDY DESIGN:
Intervention Model Description: Double-blind randomized-controlled cross-over trial consisting of two parts, including healthy adults (study part 1 - proof of concept) and adults with known diagnosis of cDI or PP (study part 2 - pilot study). Study parts 1 and 2 will be conducted consecutively. If the results of study part 1 suggest that glucagon is a potent stimulator of Copeptin in healthy adults, study part 2 will be conducted.
  The half of the study group will start with test day A (injection of glucagon), followed by test day B (injection of placebo) and the other half will start with test day B (injection of placebo), followed by test day A (injection of glucagon). The randomization will be performed by an independent third party.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study part 1: healthy adult volunteers (Experimental): 22 Healthy volunteers: The half of the study group will start with test day A (injection of glucagon), followed by test day B (injection of placebo) and the other half will start with test day B (injection of placebo), followed by test day A (injection of glucagon).
  Interventions: Diagnostic Test: Glucagon; Diagnostic Test: Placebo
- study part 2: adult patients with primary polydipsia or central diabetes insipidus (Experimental): If results of study part 1 suggest that glucagon stimulates copeptin (proof of concept),10 patients with primary polydipsia and 10 patients with central diabetes insipidus will be additionally included (study part 2): The half of the study group will start with test day A (injection of glucagon), followed by test day B (injection of placebo) and the other half will start with test day B (injection of placebo), followed by test day A (injection of glucagon).
  Interventions: Diagnostic Test: Glucagon; Diagnostic Test: Placebo

INTERVENTIONS:
Diagnostic Test: Glucagon — Glucagon with the empirical formula of C153H225N43O49S, and a molecular weight of 3483 g/mol, is a single-chain polypeptide containing 29 amino acid residues. Glucagon is provided in a single dose vial as powder. One container contains 1 mg of glucagon which results in a concentration of 1 mg/ml after dissolution in a volume of 1 ml (Glucagen NovoNordisk (Hypokit)). The currently used standard dose regimen is 1 mg of glucagon in adults. The solution for subcutaneous injection will be prepared by the study personnel according to the attached package leaflet.
Diagnostic Test: Placebo — As placebo 1 ml sodium chloride (NaCl) 0.9% to inject subcutaneous is used. It has the same optical appearance as glucagon.

SUMMARY:
This study is to evaluate copeptin values after the subcutaneous injection of glucagon in adults (healthy volunteers and patients with diabetes insipidus or primary polydipsia). It is to investigate whether glucagon stimulates the release of copeptin as a surrogate of vasopressin.

DETAILED DESCRIPTION:
The differentiation between central diabetes insipidus (cDI) and primary polydipsia (PP) is cumbersome. To date the test with the highest diagnostic accuracy is copeptin measurement after hypertonic saline Infusion.

Instead of hypertonic saline Infusion, arginine infusion - known to stimulate growth hormone - is a potent stimulator of the neurohypophysis and provides a new diagnostic tool in the differential diagnosis of cDI. Copeptin measurements upon arginine stimulation discriminated patients with diabetes insipidus vs. patients with primary polydipsia with a high diagnostic accuracy of 94%. Glucagon has been shown to stimulate GH-secretion. In analogy to the known stimulatory effect of arginine Infusion it is hypothesized that glucagon might stimulate the posterior pituitary gland and could therefore be a novel diagnostic test in the polyuria-polydipsia syndrome.

This study is to evaluate copeptin values after the subcutaneous injection of glucagon in adults (healthy volunteers and patients with diabetes insipidus or primary polydipsia).

This study is planned as a double-blind randomized-controlled cross-over trial consisting of two parts, including healthy adults (study part 1 - proof of concept) and adults with known diagnosis of cDI or PP (study part 2 - pilot study). Study parts 1 and 2 will be conducted consecutively. If the results of study part 1 suggest that glucagon is a potent stimulator of Copeptin in healthy adults, study part 2 will be conducted. Participants will receive glucagon injection and placebo injection in random order.

ELIGIBILITY:
Inclusion Criteria for healthy volunteers:

* no medication except hormonal contraception

Inclusion criteria for patients:

* Documented primary polydipsia or diabetes insipidus based on a water deprivation test or hypertonic saline Infusion
* Accordingly patients must have evidence of disordered drinking habits and diuresis defined as polyuria >50ml/kg body weight/24h and polydipsia >3l /24h, or must be on regular daily Desmopressin medication.

Exclusion Criteria for healthy volunteers:

* BMI > 25kg/m2 or < 18.5 kg/m2
* participation in a trial with investigational drugs within 30 days
* vigorous physical exercise within 24 hours before the study participation
* Alcohol intake within 24 hours before study participation
* pregnancy and breastfeeding
* Evidence of disordered drinking habits and diuresis defined as polyuria >50ml/kg Body weight/24h and polydipsia >3l /24h
* Intention to become pregnant during the study
* Known allergy towards glucagon
* Evidence of an acute illness
* Long QT syndrome
* Hemoglobin level below 120 g/l

Exclusion criteria for patients:

* BMI > 25kg/m2 or < 18.5 kg/m2
* participation in a trial with investigational drugs within 30 days
* vigorous physical exercise within 24 hours before the study participation
* Alcohol intake within 24 hours before study participation
* pregnancy and breastfeeding
* Evidence of an acute illness
* Long QT syndrome
* Hemoglobin level below 120 g/l

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Maximal increase in copeptin level | Within three hours after the injection
  Maximal increase in copeptin level within three hours after the injection of a single subcutaneous dose of 1mg glucagon or 0.9% NaCl. That is the difference between the maximal copeptin value measured between 30 and 180 minutes after the injection and the baseline value.
  measured before the injection.

SECONDARY OUTCOMES:
Change in copeptin values | Measured at 0 (baseline), 30, 60, 90, 120, 150 and 180 minutes after injection
  Change in copeptin values
Maximum copeptin time: the time from baseline to the maximum copeptin value | Within three hours after the injection
  Maximum copeptin time: the time from baseline to the maximum copeptin value
Change in growth hormone (GH) | Measured at 0 (baseline), 30, 60, 90, 120, 150 and 180 minutes after injection
  Change in growth hormone (GH)
Change in prolactin | Measured at 0 (baseline), 30, 60, 90, 120, 150 and 180 minutes after injection
  Change in prolactin
Change in plasma sodium | Measured at 0 (baseline), 30, 60, 90, 120, 150 and 180 minutes after injection
  Change in plasma sodium
Change in plasma osmolality | Measured at 0 (baseline), 30, 60, 90, 120, 150 and 180 minutes after injection
  Change in plasma osmolality
Change in oxytocin | Measured at 0 (baseline), 30, 60, 90, 120, 150 and 180 minutes after injection
  Change in oxytocin
Maximal Change in GH | Within three hours after the injection
  Maximal Change in GH
Maximal Change in prolactin | Within three hours after the injection
  Maximal Change in prolactin
Maximal Change in plasma osmolality | Within three hours after the injection
  Maximal Change in plasma osmolality
Maximal Change in oxytocin | Within three hours after the injection
  Maximal Change in oxytocin

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr. med., Principal Investigator — Endocrinology, Diabetes and Metabolism, University Hospital Basel
Locations (1):
- Divison of Endocrinology, Diabetes and Metabolism,University Hospital Basel, Basel, Switzerland